CLINICAL TRIAL: NCT01307189
Title: Effects of Tiotropium on Walking Capacity in Patients With COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Dr François Maltals, Laval University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CER1199
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Exercise; Endurance shuttle walking test; Bronchodilation; Tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tiotropium (Active Comparator)
  Interventions: Drug: Tiotropium
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiotropium — Tiotropium diskus inhalation powder, 18ug, once daily
  Other Names: Spiriva
  Arms: Tiotropium
Drug: Placebo — Placebo diskus inhalation powder, once daily
  Arms: Placebo

SUMMARY:
This study was designed to test the following hypothesis:

A) The acute and long-term (3 weeks) bronchodilator-induced changes in exercise tolerance and in the physiological response during the endurance shuttle walk will be greater with tiotropium compared to placebo in COPD patients.

B) Three weeks of bronchodilation will be associated with increase activity of daily living as evaluated using the London Chest Activity Daily Living scale.

DETAILED DESCRIPTION:
Objectives:

The purpose of this study is to compare the acute bronchodilator-induced changes in exercise tolerance during the endurance shuttle walk between tiotropium and placebo in COPD patients. Also, it will evaluate the physiological response (VE, VO2, VCO2, and heart rate) during the endurance shuttle walk in patients with COPD patients. Finally, it will compare the long-term (3 weeks) bronchodilator-induced changes in exercise tolerance during the endurance shuttle walk between tiotropium and placebo in COPD patients and evaluate the impact of long-term (3 weeks) bronchodilation on activity of daily living evaluated using the London Chest Activity Daily Living scale.

Methods:

This will be a double-blind, randomized and parallel-group study. Due to the long action duration of tiotropium (up to 4 weeks), a cross-over design, as we used in our ipratropium versus placebo study, is not appropriate in the present study. The study will require five visits at the Centre de recherche de l'Hopital Laval. The first visit will include review of the consent form, pulmonary function testing, and a maximal incremental shuttle walk. The following two visits (Visit 2 and 3) will be used to familiarize the participants to the shuttle endurance walking test. Salbutamol and ipratropium bromide will be stopped 6 hours prior to these visits while the remaining medication allowed during the study period (see below) will be continued as prescribed. The goal of the familiarization will be to reduce the learning effect that typically occurs when an individual completes the same endurance test several times 3. On visit 4, patients will be randomized to receive one of the two treatments: placebo or tiotropium 18 ug (Spiriva) using the handihaler device. Pulmonary function testing will then be performed and the London Chest Activity Daily Living scale will be administered. Two hours following the inhalation of the first study dose, pulmonary function testing will be repeated and the patients will perform an endurance shuttle walk. They will be provided enough medication for the study duration and discharged. The same procedure as Visit 4 will be completed three weeks later, on visit 5.

Data analysis:

The main outcome will be endurance time at day 21. This variable will be compared between the two treatment arms using an unpaired t-test. The endurance time at day 0 will also be compared between the two treatment arms using the same procedure. The time course of the cardiorespiratory parameters and dyspnea over time will be compared between the two exercise modalities. Comparisons will be done using a repeated measure design (ANOVA). Significance level will be set at a p value of 0.05. The two familiarization endurance shuttle walk tests performed at day -10 and day -5 will be used to evaluate the test-retest variability of this procedure.

ELIGIBILITY:
Inclusion Criteria:

* age > 50 years, smoking history > 10 packs/year, FEV1 < 70% of predicted and FEV1/FVC < 70%.

Exclusion Criteria:

* respiratory exacerbation within the 2 months preceding the study, history of asthma, significant O2 desaturation (SaO2 < 85%) at rest or during exercise, presence of another pathology that could influence exercise tolerance.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-04; Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Endurance time during an endurance shuttle walk | acute response (2.5 hours) following the administration of the active and comparison drug

SECONDARY OUTCOMES:
Compare the long-term bronchodilator-induced changes in exercise tolerance during the endurance shuttle walk | three weeks
Evaluate the impact of long-term bronchodilation on activity of daily living evaluated using the London Chest Activity Daily Living scale | three weeks
Cardio-respiratory responses during an endurance shutlle walk | acute response following the administration of the study medication

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Principal Investigator — Laval University
Locations (1):
- Centre de recherche de l'IUCPQ, Québec, Quebec, Canada